CLINICAL TRIAL: NCT06601491
Title: Lifestyle Randomised Intervention for Healthy Vascular Ageing - a Multifactorial Assessment of Vascular Ageing Among Cypriots in Early Adulthood Through Biobank.cy
Brief Title: Early Vascular Ageing Among Cypriots
Acronym: LifeEVA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cyprus (Other)
Collaborators: Aristotle University Of Thessaloniki (Other); Harokopio University (Other)
Responsible Party: Principal Investigator, Panagiota Veloudi, Researcher, University of Cyprus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EEBK/2024/21
Record Dates: First submitted 2024-08-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Vascular Stiffness; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Lifestyle Intervention
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Lifestyle Intervention — Participants in the intervention group receive structured, pesonalised lifestyle, dietary and physical activity consultations. They undergo various assessments such as aortic stiffness measurement, blood pressure measurement, and complete several questionnaires (e.g., whole exome sequencing, IPAQ, handgrip strength, socio-demographic, clinical history, quality of life, smoking, alcohol consumption, sleep patterns, stress assessment).
  Arms: Intervention

SUMMARY:
The LifeEVA project aims to tackle the significant public health challenge of cardiovascular disease (CVD) by addressing early vascular ageing (EVA), characterized by increased arterial stiffness and reduced vascular compliance, particularly in young adults. The project seeks to develop and implement innovative, personalized lifestyle interventions targeting Cypriots aged 18-40 who are overweight or obese. Utilizing genetic data from biobank.cy, LifeEVA aims to understand the progression of EVA and reduce CVD risk through tailored dietary and physical activity counseling.

The methodology involves a prospective, randomized, open-label, blinded endpoint trial over one year. Participants will be recruited from biobank.cy's database, ensuring a robust sample. They will receive personalized interventions based on their genetic profile, including a hypocaloric diet, physical activity plan and taking into account other factors (i.e. sleep, anxiety etc). The project's work is divided into five work packages: project management, dissemination and exploitation activities, baseline assessment and recruitment, intervention implementation and data collection, and data analysis and manuscript preparation.

Anticipated results include significant reductions in vascular stiffness, improved cardiovascular health markers, and enhanced understanding of the interplay between genetics and lifestyle in EVA. The project's impact extends to the establishment of a vascular health assessment clinic, contributions to public health by reducing CVD prevalence, and advancing the field of personalized preventive healthcare. LifeEVA is positioned to make significant contributions to cardiovascular research, promote innovation, and enhance the scientific and public health landscape in Cyprus.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 40 years old.
* BMI≥25 kg/m².
* WC≥0.9 m for men and ≥0.8 m for women

Exclusion Criteria:

* Individuals with a history of eating disorders.
* Those with significant chronic diseases like advanced cardiovascular diseases
* Pregnant or breastfeeding women or women to intend/are in the process of trying to get pregnant within 1-year after intervention onset.
* Individuals currently on medication or diets that significantly affect metabolism or body weight.
* Those who have participated in another weight loss program or study within the last six months.
* Taking any vasoactive medications.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 352 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Vascular Stiffness as Measured Through Pulse Wave Velocity at 12 Months | Every three months, duration: 1 year
  Vascular stiffness will be assessed by measuring pulse wave velocity. Pulse wave velocity is the speed at which the arterial pulse travels through the circulatory system, a key indicator of arterial stiffness.

CONTACTS AND LOCATIONS:
Overall Officials: Panagiota Veloudi, PhD, Principal Investigator — University of Cyprus; Eleni M Loizidou, PhD, Principal Investigator — Cyprus Institute of Neurology and Genetics; Constantinos Deltas, PhD, Principal Investigator — University of Cyprus
Locations (1):
- biobank.cy Center of Excellence in Biobanking and Biomedical Research, University of Cyprus, Nicosia, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No